CLINICAL TRIAL: NCT06392919
Title: Effects of Perioperative Repetitive Transcranial Magnetic Stimulation on Postoperative Delirium, Postoperative Cognitive Dysfunction, and Chronic Post-surgical Pain in Elderly Surgical Patients
Brief Title: The Impact of Repetitive Transcranial Magnetic Stimulation on the Prognosis of Elderly Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Chaochao Zhong, Principal Investigator, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-K005-01
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction; Chronic Post-surgical Pain
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Pain, Postoperative | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham repetitive transcranial magnetic stimulation (rTMS group) (No Intervention): After the surgical anesthesia, the patient is transferred to the Post-Anesthesia Care Unit (PACU). The Sham rTMS intervention occurs after the tracheal tube is removed in the PACU.In the sham rTMS group, the setup, including the stimulation site and parameters, is identical to that of the rTMS group. However, although the rTMS device is connected to the patient, no actual stimulation is delivered.
- repetitive transcranial magnetic stimulation (rTMS group) (Experimental): After the surgical anesthesia, the patient is transferred to the Post-Anesthesia Care Unit (PACU). The rTMS intervention occurs after the tracheal tube is removed in the PACU. The stimulation site is the DLPFC (left dorsolateral prefrontal cortex); the stimulation intensity is 100% of the Resting Motor Threshold (RMT); the frequency is 10 Hz; and the total number of pulses is 2000. The pulse characteristics include a duration of 5 seconds per session with a 25-second interval between sessions.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS intervention timing: rTMS is applied after the tracheal tube is removed in the PACU. Stimulation site: DLPFC (left dorsolateral prefrontal cortex); Stimulation intensity: 100% RMT; Stimulation frequency: 10Hz; Total number of stimulation pulses: 2000. Pulse characteristics: Each duration lasts 5 seconds, with a 25-second interval.
  Arms: repetitive transcranial magnetic stimulation (rTMS group)

SUMMARY:
Exploring the effects of repeated transcranial magnetic stimulation (rTMS) during the perioperative period on the incidence of postoperative delirium, postoperative cognitive dysfunction, and chronic postoperative pain in elderly patients, as well as its possible mechanisms.

DETAILED DESCRIPTION:
Patients are recruited one week prior to the trial commencement, during which they are informed about the experimental protocol and associated risks. After obtaining informed consent and signatures, they are enrolled as study participants.Patients who meet the trial criteria are randomly assigned in a 1:1 ratio to the control group (sham rTMS group) and the intervention group (rTMS group, with rTMS intervention applied in the PACU after surgery) in a double-blind manner (with rTMS intervention and postoperative follow-up conducted by different researchers).

Note: This trial includes three co-primary outcomes-postoperative delirium (POD), postoperative cognitive dysfunction (POCD), and chronic postoperative pain (CPSP). To account for the different nature and timelines of these outcomes, the study was designed to include two parallel patient cohorts under a unified protocol:

1. Elderly patients undergoing gastrointestinal surgery are enrolled primarily for the evaluation of POD, a short-term outcome assessed within 3 days postoperatively.
2. Elderly patients undergoing thoracic surgery are enrolled to evaluate POCD (at 1 month) and CPSP (at 3 months), which are longer-term outcomes.

These two patient cohorts are studied concurrently but analyzed separately according to outcome-specific follow-up timelines and sample size estimations. A total of 122 gastrointestinal surgery patients were enrolled and analyzed for POD. The maximum estimated sample size is for the POCD and CPSP cohort (n=230). Results will be reported in phases corresponding to the completion of each outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;
* ASA ≤ 3;
* Elective surgery patients.

Exclusion Criteria:

* Refusal to sign the consent form;
* Mini-Mental State Examination (MMSE) score < 15;
* Preoperative neuropsychiatric diseases and history of neurological or psychiatric disorders;
* Preoperative cranial or scalp injuries;
* History of drug or alcohol abuse; Visual or auditory impairments, communication difficulties; Presence of metallic implants in the body; Preoperative history of severe cardiovascular disease or severe liver or kidney dysfunction.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium during the first 3 days after surgery | The first 3 days after surgery
  Delirium is assessed twice daily (8-10 AM and 6-8 PM) with the Confusion Assessment Method for patients without endotracheal intubation during the first 3 days after surgery.
Incidence of Postoperative Cognitive Dysfunction | 1 month after surgery
  Cognitive function assessed with MoCA (Montreal Cognitive Assessment) test on the 30th day after surgery
Incidence of chronic postsurgical pain (CPSP) at 3 months after surgery | At 3 months after surgery
  CPSP is defined as pain persisting for at least three months after surgery that was not present before surgery or that had different characteristics, and other possible causes of pain were excluded (e.g., cancer recurrence, infection). Pain intensity is assessed with the numeric rating scale, an 11-point scale where 0=no pain and 10=the worst pain, both at rest and with movement.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chao Zhong, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No